CLINICAL TRIAL: NCT05317286
Title: Prospective Validation of a Deep Learning Algorithm for Prediction of the Left Ventricular Ejection Fraction From Coronary Angiogram Videos in Patients With Acute Coronary Syndrome
Brief Title: LVEF Prediction During ACS Using AI Algorithm Applied on Coronary Angiogram Videos
Acronym: CathEF
Status: Completed | Type: Observational
Sponsor: Montreal Heart Institute (Other)
Collaborators: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Robert Avram, Principal Investigator, Montreal Heart Institute
Other Study IDs: CathEF
Record Dates: First submitted 2022-03-22; First posted 2022-04-07 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Acute Coronary Syndrome; Left Ventricular Dysfunction
Keywords: acute coronary syndrome; coronary angiogram; left ventricular ejection fraction; ventriculography; artificial intelligence
MeSH Terms: conditions — Acute Coronary Syndrome; Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Left ventricular ejection fraction (LVEF) is one of the strongest predictors of mortality and morbidity in patients with acute coronary syndrome (ACS). Transthoracic echocardiography (TTE) remains the gold standard for LVEF measurement. Currently, LVEF can be estimated at the time of the coronary angiogram but requires a ventriculography. This latter is performed at the price of an increased amount of contrast media injected and puts the patients at risk for mechanical complications, ventricular arrhythmia or atrio-ventricular blocks. Artificial intelligence (AI) has previously been shown to be an accurate method for determining LVEF using different data sources. Fur the purpose of this study, we aim at validating prospectively an AI algorithm, called CathEF, for the prediction of real-time LVEF (AI-LVEF) compared to TTE-LVEF and ventriculography in patients undergoing coronary angiogram for ACS.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed by the participant
* Acute coronary syndrome
* Creatinine clearance ≥30 ml/min/m2 according to MDRD

Exclusion Criteria:

* Creatinine clearance <30 ml/min/m2 according to MDRD
* No indication to perform TTE in the 7 days following coronary angiogram
* Right bundle branch block
* Suspected or confirmed left ventricular thrombus
* Suspected or confirmed aortic dissection
* Ventriculography not feasible
* No left coronary system angiogram

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults treated by percutaneous coronary intervention for ACS in whom left ventriculography is not contra-indicated and TTE-LVEF is expected to be measured in the next 24h to 7 days.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Area under the curve-Receiver Operating Characteristics (AUC-ROC) of the CathEF algorithm for differentiating a LVEF ≤ or >50%, compared to TTE-LVEF | Either 7 days before or up to 7 days after the coronary angiogram

SECONDARY OUTCOMES:
Comparing AUC-ROC of CathEF and ventriculography for differentiating a LVEF ≤ or >50% | Either 7 days before or up to 7 days after the coronary angiogram
Sensitivity of CathEF and ventriculography for differentiating a LVEF ≤ or >50% in comparison to TTE-LVEF. | Either 7 days before or up to 7 days after the coronary angiogram
Specificity of CathEF and ventriculography for differentiating a LVEF ≤ or >50% in comparison to TTE-LVEF. | Either 7 days before or up to 7 days after the coronary angiogram
Number of participants with major adverse cardiovascular events (Combined outcome of combined outcomeof mortality, ventricular arrhythmia requiring an intervention, heart failure, need for inotropic support, renal failure KDIGO≥2 and stroke) | At 7 days or before discharge, if earlier.
AUC-ROC of the re-trained CathEF algorthim for differentiating a LEVF ≤ or >50% | Either 7 days before or up to 7 days after the coronary angiogram
Sensitivity of the re-trained CathEF algorthim for differentiating a LEVF ≤ or >50% | Either 7 days before or up to 7 days after the coronary angiogram
Specificity of the re-trained CathEF algorthim for differentiating a LEVF ≤ or >50% | Either 7 days before or up to 7 days after the coronary angiogram
Likert scale on the impact on the procedure, ease of use and utility of the CathEF algorithm in the clinical practice, as assessed by interventional cardiologists | Through study completion, an average of 1 year.

CONTACTS AND LOCATIONS:
Locations (1):
- Robert Avram, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared to other researchers on reasonable request to the principal investigator.